CLINICAL TRIAL: NCT01959412
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Crossover Study to Evaluate the Efficacy, Safety and Tolerability of Five Different Doses of Inhaled Indacaterol (QAB149) Delivered Via the Single Dose Dry Powder Inhaler (SDDPI) in Patients With Persistent Asthma
Brief Title: Crossover Study to Evaluate the Efficacy, Safety and Tolerability of Different Doses of Indacaterol in Patients With Persistent Asthma
Acronym: QAB149
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CQVA149A2210
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Results first posted 2015-05-06 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-04

CONDITIONS: Asthma
Keywords: wheezing, short of breath, laba, inhaler
MeSH Terms: conditions — Asthma; Respiratory Sounds; Dyspnea | interventions — indacaterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Treatment Period Sequence 1 (Experimental): Indacaterol 37.5 mcg in the morning + matching placebo in the evening, 14 days later indacaterol 55 mcg in the morning + matching placebo in the evening, 14 days later placebo in the morning + matching placebo in the evening, 14 days later indacaterol 75 mcg in the morning + matching placebo in the evening, 14 days later indacaterol 27.5 mcg in the morning + 27.5 mcgin the evening, 14 days later indacaterol 150 mcg in the morning + matching placebo in the evening
  Interventions: Drug: Indacaterol 27.5 mcg; Drug: Placebo
- Treatment Period Sequence 2 (Experimental): Indacaterol 55 mcg in the morning + matching placebo in the evening, 14 days later indacaterol 75 mcg in the morning + matching placebo in the evening, 14 days later 37.5 in the morning + matching placebo in the evening, 14 days later indacaterol 150 mcg in the morning + matching placebo in the evening, 14 days later placebo in the morning + placebo in the evening, 14 days later indacaterol 27.5 mcg in the morning + 27.5 mcg in the evening
  Interventions: Drug: Indacaterol 37.5; Drug: Placebo
- Treatment Period Sequence 3 (Experimental): Indacaterol 75 mcg in the morning + matching placebo in the evening, 14 days later indacaterol 150 mcg in the morning + matching placebo in the evening, 14 days later 55mcg in the morning + matching placebo in the evening, 14 days later indacaterol 27.5 mcg in the morning + 27.5 mcg in the evening, 14 days later indacaterol 37.5 mcg in the morning + matching placebo n the evening, 14 days later placebo in the morning + matching placebo in the evening
  Interventions: Drug: Indacaterol 55 mcg; Drug: Placebo
- Treatment Sequence Period 4 (Experimental): Indacaterol 150 mcg in the morning + matching placebo in the evening, 14 days later indacaterol 27.5 mcg in the morning + 27.5 mcg in the evening, 14 days later 75 mcg in the morning + matching placebo in the evening, 14 days later placebo in the morning + matching placebo in the evening, 14 days later indacaterol 55 mcg in the morning + matching placebo in the evening, 14 days later indacaterol 37.5 mcg in the morning + matching placebo in the evening
  Interventions: Drug: Indacaterol 75 mcg; Drug: Placebo
- Treatment Period Sequence 5 (Experimental): Indacaterol 27.5 mcg in the morning + 27.5mcg in the evening, 14 days later placebo in the morning + matching placebo in the evening, 14 days later 150mcg in the morning + matching placebo in the evening, 14 days later indacaterol 37.5 mcg in the morning + matching placebo in the evening, 14 days later indacaterol 75 mcg in the morning + matching placebo in the evening, 14 days later indacaterol 55 mcg in the morning + matching placebo in the evening
  Interventions: Drug: Indacaterol 150 mcg; Drug: Placebo
- Treatment Period Sequence 6 (Experimental): Placebo in the morning + matching placebo in the evening, 14 days later indacaterol 37.5 mcg in the morning + matching placebo in the evening, 14 days later 27.5 mcg in the morning + 27.5mcg in the evening, 14 days later indacaterol 55 mcg in the morning + matching placebo in the evening, 14 days later indacaterol 150 mcg in the morning + matching placebo in the evening, 14 days later 75 mcg in the morning + matching placebo in the evening
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Indacaterol 27.5 mcg — indacaterol 27.5 mcg twice daily inhaled once via inhaler
  Arms: Treatment Period Sequence 1
Drug: Indacaterol 37.5 — Indacaterol 37.5 mcg once daily, inhaled once via inhaler
  Arms: Treatment Period Sequence 2
Drug: Indacaterol 55 mcg — Indacaterol 55 mcg once daily, inhaled once via inhaler
  Arms: Treatment Period Sequence 3
Drug: Indacaterol 75 mcg — Indacaterol 75 mcg once daily, inhaled once via inhaler
  Arms: Treatment Sequence Period 4
Drug: Indacaterol 150 mcg — Indacaterol 150 mcg once daily, inhaled once via inhaler
  Arms: Treatment Period Sequence 5
Drug: Placebo — Placebo to indacaterol once or twice daily (depending on assigned sequence) via inlaher

SUMMARY:
The purpose of this study is to determine the efficacy of indacaterol 55µg once daily (and 27.5 µg twice) in QVA149 compared to 75 µg indacaterol monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Asthma for at least 6 months, using inhaled corticosteroid for at least one month, foreced breath test less than below the normal value of the general population, -show an immediate improvement in breathing when given albuterol

Exclusion Criteria:

* patients who have smoked in the past 6 months or are currently smoking, including those who smoked more than a pack of cigarettes a day for at least 10 years, -patients who have a history of life-threatening asthma, -patients who have had an astham attack, in the last 6 weeks, requiring use of systemic steroids, hospitalization, or ER visit, -patients who have had a respiratory tract infection or worsening asthma between screening or run-in periods, patients requring use of other asthma-related drugs during the trial, other protocol-defined inclusion/exclusion may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2013-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- United States (12):
  - Novartis Investigative Site, Huntington Beach, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Mission Viejo, California
  - Novartis Investigative Site, Centennial, Colorado
  - Novartis Investigative Site, North Dartmouth, Massachusetts
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Skillman, New Jersey
  - Novartis Investigative Site, Raleigh, North Carolina
  - Novartis Investigative Site, Medford, Oregon
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, El Paso, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 4 (Ind 150 μg): indacaterol 150 μg, indacaterol 27.5 μg, indacaterol 75 μg, placebo indacaterol 55 μg indacaterol 37.5 μg Indacaterol 150 mcg in the morning + matching placebo in the evening, 14 days later indacaterol 27.5 mcg in the morning + 27.5 mcg in the evening, 14 days later 75 mcg in the morning + matching placebo in the evening, 14 days later placebo in the morning + matching placebo in the evening, 14 days later indacaterol 55 mcg in the morning + matching placebo in the evening, 14 days later indacaterol 37.5 mcg in the morning + matching placebo in the evening
- Sequence 3 (Ind 75 μg): indacaterol 75 μg indacaterol 150 μg indacaterol 55 μg indacaterol 27.5 μg indacaterol 37.5 μg placebo Indacaterol 75 mcg in the morning + matching placebo in the evening, 14 days later indacaterol 150 mcg in the morning + matching placebo in the evening, 14 days later 55mcg in the morning + matching placebo in the evening, 14 days later indacaterol 27.5 mcg in the morning + 27.5 mcg in the evening, 14 days later indacaterol 37.5 mcg in the morning + matching placebo n the evening, 14 days later placebo in the morning + matching placebo in the evening
- Sequence 2 (Ind 55 μg): indacaterol 55 μg indacaterol 75 μg indacaterol 37.5 μg indacaterol 150 μg placebo indacaterol 27.5 μg Indacaterol 55 mcg in the morning + matching placebo in the evening, 14 days later indacaterol 75 mcg in the morning + matching placebo in the evening, 14 days later 37.5 in the morning + matching placebo in the evening, 14 days later indacaterol 150 mcg in the morning + matching placebo in the evening, 14 days later placebo in the morning + placebo in the evening, 14 days later indacaterol 27.5 mcg in the morning + 27.5 mcg in the evening
- Sequence 1 (Ind 37.5 μg): indacaterol 37.5 μg indacaterol 55μg Placebo indacaterol 75μg indacaterol 27.5μg indacaterol 150μg indacaterol 37.5 mcg in the morning + matching placebo in the evening, 14 days later indacaterol 55 mcg in the morning + matching placebo in the evening, 14 days later placebo in the morning + matching placebo in the evening, 14 days later indacaterol 75 mcg in the morning + matching placebo in the evening, 14 days later indacaterol 27.5 mcg in the morning + 27.5 mcgin the evening, 14 days later indacaterol 150 mcg in the morning + matching placebo in the evening
- Sequence 5 (Ind 27.5 μg): indacaterol 27.5 μg placebo indacaterol 150 μg indacaterol 37.5 μg indacaterol 75 μg indacaterol 55 μg Indacaterol 27.5 mcg in the morning + 27.5mcg in the evening, 14 days later placebo in the morning + matching placebo in the evening, 14 days later 150mcg in the morning + matching placebo in the evening, 14 days later indacaterol 37.5 mcg in the morning + matching placebo in the evening, 14 days later indacaterol 75 mcg in the morning + matching placebo in the evening, 14 days later indacaterol 55 mcg in the morning + matching placebo in the evening
- Sequence 6 (Placebo): Placebo, indacaterol 37.5 μg, indacaterol 27.5 μg indacaterol 55 μg, indacaterol 150 μg, indacaterol 75 μg Placebo in the morning + matching placebo in the evening, 14 days later indacaterol 37.5 mcg in the morning + matching placebo in the evening, 14 days later 27.5 mcg in the morning + 27.5mcg in the evening, 14 days later indacaterol 55 mcg in the morning + matching placebo in the evening, 14 days later indacaterol 150 mcg in the morning + matching placebo in the evening, 14 days later 75 mcg in the morning + matching placebo in the evening
Period: Overall Study
Arm/Group | Sequence 4 (Ind 150 μg) | Sequence 3 (Ind 75 μg) | Sequence 2 (Ind 55 μg) | Sequence 1 (Ind 37.5 μg) | Sequence 5 (Ind 27.5 μg) | Sequence 6 (Placebo)
Started | 15 | 15 | 15 | 15 | 16 | 15
Completed | 14 | 14 | 15 | 13 | 13 | 15
Not Completed | 1 | 1 | 0 | 2 | 3 | 0
Not completed — Protocol deviation | 1 | 1 | 0 | 1 | 3 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants randomized to one of six treatment sequences
Arm/Group | All Participants
Number analyzed (Participants) | 91
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.4 (13.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 38

OUTCOME MEASURES:

1. Primary Outcome: Change From Period Baseline in FEV1 (L) AUC(0-24h)
Description: Forced Expiratory Volume in 1 second (FEV1) is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. FEV1 will be measured pre-dose and over a 24 hours post-dose period.
Time Frame: Day 1 (24 hours)
Population: drug. Following the intent-to-treat principle, data for patients in the FAS were analyzed according to the treatment they were randomized to in the assigned treatment sequence. The FAS was used in the analysis of all efficacy variables
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- Ind 150 μg: Indacaterol 150 mcg in the morning + matching placebo in the evening, 14 days later indacaterol 27.5 mcg in the morning + 27.5 mcg in the evening, 14 days later 75 mcg in the morning + matching placebo in the evening, 14 days later placebo in the morning + matching placebo in the evening, 14 days later indacaterol 55 mcg in the morning + matching placebo in the evening, 14 days later indacaterol 37.5 mcg in the morning + matching placebo in the evening
- Ind 75 μg: Indacaterol 75 mcg in the morning + matching placebo in the evening, 14 days later indacaterol 150 mcg in the morning + matching placebo in the evening, 14 days later 55mcg in the morning + matching placebo in the evening, 14 days later indacaterol 27.5 mcg in the morning + 27.5 mcg in the evening, 14 days later indacaterol 37.5 mcg in the morning + matching placebo n the evening, 14 days later placebo in the morning + matching placebo in the evening
- Ind 55 μg: Indacaterol 55 mcg in the morning + matching placebo in the evening, 14 days later indacaterol 75 mcg in the morning + matching placebo in the evening, 14 days later 37.5 in the morning + matching placebo in the evening, 14 days later indacaterol 150 mcg in the morning + matching placebo in the evening, 14 days later placebo in the morning + placebo in the evening, 14 days later indacaterol 27.5 mcg in the morning + 27.5 mcg in the evening
- Ind 37.5 μg: Indacaterol 37.5 mcg in the morning + matching placebo in the evening, 14 days later indacaterol 55 mcg in the morning + matching placebo in the evening, 14 days later placebo in the morning + matching placebo in the evening, 14 days later indacaterol 75 mcg in the morning + matching placebo in the evening, 14 days later indacaterol 27.5 mcg in the morning + 27.5 mcgin the evening, 14 days later indacaterol 150 mcg in the morning + matching placebo in the evening
- Ind 27.5: Indacaterol 27.5 mcg in the morning + 27.5mcg in the evening, 14 days later placebo in the morning + matching placebo in the evening, 14 days later 150mcg in the morning + matching placebo in the evening, 14 days later indacaterol 37.5 mcg in the morning + matching placebo in the evening, 14 days later indacaterol 75 mcg in the morning + matching placebo in the evening, 14 days later indacaterol 55 mcg in the morning + matching placebo in the evening
- Placebo: Placebo in the morning + matching placebo in the evening, 14 days later indacaterol 37.5 mcg in the morning + matching placebo in the evening, 14 days later 27.5 mcg in the morning + 27.5mcg in the evening, 14 days later indacaterol 55 mcg in the morning + matching placebo in the evening, 14 days later indacaterol 150 mcg in the morning + matching placebo in the evening, 14 days later 75 mcg in the morning + matching placebo in the evening
Arm/Group | Ind 150 μg | Ind 75 μg | Ind 55 μg | Ind 37.5 μg | Ind 27.5 | Placebo
Number analyzed (Participants) | 84 | 86 | 85 | 84 | 87 | 86
Liters | 0.209 (0.0153) | 0.165 (0.0152) | 0.154 (0.0152) | 0.121 (0.0153) | 0.143 (0.0151) | 0.022 (0.0152)

2. Secondary Outcome: Change From Period Baseline in FEV1 (L) AUC(0-12h) and FEV1 (L) AUC(12- 24h)
Description: Forced Expiratory Volume in 1 second (FEV1) is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. FEV1 will be measured pre-dose and over a 12 hours post-dose period.
Time Frame: Day 1 (12 hours)
Population: The Full Analysis Set (FAS) consisted of all patients in the RAN who received at least 1 dose of study drug. Following the intent-to-treat principle, data for patients in the FAS were analyzed according to the treatment they were randomized to in the assigned treatment sequence. The FAS was used in the analysis of all efficacy variables
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Ind 150 μg | Ind 75 μg | Ind 55 μg | Ind 37.5 μg | Ind 27.5 | Placebo
Number analyzed (Participants) | 84 | 86 | 85 | 84 | 87 | 86
liters
  FEV1 AUC (0-12h) | 0.229 (0.0150) | 0.180 (0.0148) | 0.176 (0.0149) | 0.131 (0.0150) | 0.125 (0.0148) | 0.036 (0.0148)
  FEV1 AUC (12-24h) | 0.190 (0.0177) | 0.153 (0.0175) | 0.136 (0.0176) | 0.115 (0.0177) | 0.164 (0.0175) | 0.012 (0.0175)

3. Secondary Outcome: Change From Period Baseline in Peak FEV1 (L)
Description: Spirometry will be conducted according to internationally accepted standards. Peak Forced Expiratory Volume in 1 second (FEV1) is the maximum FEV1 recorded between different time points.
Time Frame: Day 1 (24 hours)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Ind 150 μg | Ind 75 μg | Ind 55 μg | Ind 37.5 μg | Ind 27.5 | Placebo
Number analyzed (Participants) | 84 | 86 | 85 | 84 | 87 | 86
Liters | 0.347 (0.0154) | 0.290 (0.0152) | 0.298 (0.0153) | 0.249 (0.0154) | 0.259 (0.0152) | 0.158 (0.0152)

4. Secondary Outcome: Change From Period Baseline in Trough FEV1 (L)
Description: Forced Expiratory Volume in 1 second (FEV1) is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation, measured through spirometry testing. The trough in FEV1 is defined as the mean of two measurements at different time points.
Time Frame: Day 1 (24 hours)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Ind 150 μg | Ind 75 μg | Ind 55 μg | Ind 37.5 μg | Ind 27.5 | Placebo
Number analyzed (Participants) | 82 | 86 | 84 | 83 | 86 | 86
Liters | 0.207 (0.0183) | 0.162 (0.0180) | 0.137 (0.0181) | 0.128 (0.0182) | 0.161 (0.0180) | 0.024 (0.0180)

5. Secondary Outcome: Change From Period Baseline in FVC (L) AUC (0-24h)
Description: Forced Vital Capacity (FVC) is the amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. FVC will be assessed via spirometry. A positive change from baseline in FVC indicates improvement in lung function.
Time Frame: Day 1 (24 hours)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Ind 150 μg | Ind 75 μg | Ind 55 μg | Ind 37.5 μg | Ind 27.5 | Placebo
Number analyzed (Participants) | 84 | 86 | 85 | 84 | 87 | 86
Liters | 0.147 (0.0183) | 0.120 (0.0181) | 0.118 (0.0182) | 0.085 (0.0183) | 0.106 (0.0180) | 0.016 (0.0181)

ADVERSE EVENTS:
Arm/Group | Ind 150 μg | Ind 75 μg | Ind 55 μg | Ind 37.5 μg | Ind 27.5 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/88 | 1/87 | 1/86 | 1/85 | 0/90 | 0/88
Other Adverse Events (participants affected / at risk) | 15/88 | 14/87 | 10/86 | 11/85 | 12/90 | 9/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ind 150 μg (N=88) | Ind 75 μg (N=87) | Ind 55 μg (N=86) | Ind 37.5 μg (N=85) | Ind 27.5 (N=90) | Placebo (N=88)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ind 150 μg (N=88) | Ind 75 μg (N=87) | Ind 55 μg (N=86) | Ind 37.5 μg (N=85) | Ind 27.5 (N=90) | Placebo (N=88)
TOOTHACHE (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
NASOPHARYNGITIS (Infections and infestations) | 2 | 3 | 0 | 0 | 0 | 2
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1 | 1 | 1 | 2 | 2
INAPPROPRIATE SCHEDULE OF DRUG ADMINISTRATION (Injury, poisoning and procedural complications) | 5 | 2 | 2 | 2 | 4 | 3
COUGH (Respiratory, thoracic and mediastinal disorders) | 8 | 8 | 5 | 8 | 6 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety